CLINICAL TRIAL: NCT07049575
Title: A Maximal Use Trial of Ruxolitinib Cream in Adult and Adolescent Participants With Hidradenitis Suppurativa
Brief Title: Study to Evaluate the Maximal Use of Ruxolitinib Cream in Adult and Adolescent Participants With Hidradenitis Suppurativa
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB018424-112
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis suppurativa; skin disease; ruxolitinb cream
MeSH Terms: conditions — Hidradenitis Suppurativa; Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib 1.5 % Cream (Experimental): Participants received ruxolitinib 1.5% cream, applied topically to the affected area as defined in the protocol.
  Interventions: Drug: Ruxolitinib Cream

INTERVENTIONS:
Drug: Ruxolitinib Cream — Ruxolitinib cream applied topically to the affected area as a thin film twice daily.

SUMMARY:
The purpose of this study is to evaluate the maximal use of ruxolitinib cream in adult and adolescent participants with hidradenitis suppurativa.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HS for at least 6 months before screening visit.
* Diagnosis of HS (Hurley Stage I, II, III) with a total abscess and inflammatory nodule count of at least 4 and affecting at least 3 distinct anatomical areas at screening and Day 1 visits.
* Total estimated treatment BSA > 20% at screening and baseline.
* Agreement to not use topical or systemic antibiotics for treatment of HS during the Maximal Use Treatment Period.
* Willingness to avoid pregnancy or fathering children based on the criteria defined in the protocol.
* Further inclusion criteria apply.

Exclusion Criteria:

* Current or history of skin condition(s) other than HS that might confound the evaluation of HS; clinically uncontrolled cardiovascular disease; thrombosis; certain cancers; certain infections; severe anemia, thrombocytopenia, or neutropenia; other medical conditions at the discretion of the investigator.
* Laboratory values outside of the protocol-defined ranges.
* Further exclusion criteria apply.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-12-09 (Estimated); Study Completion 2026-12-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 24 weeks
  Defined as adverse events reported for the first time or worsening of a pre-existing event after the first application of study drug.
Number of participants with TEAEs leading to treatment interruption, discontinuation | Up to 24 weeks
  Number of participants with TEAEs leading to dose interruption or discontinuation

SECONDARY OUTCOMES:
Pharmacokinetics Parameter (PK): Cmax of INCB018424 | Up to 24 weeks
  Defined as maximum observed plasma concentration of INCB018424.
Pharmacokinetics Parameter: Tmax of INCB018424 | Up to 24 weeks
  Defined as the time to reach the maximum plasma concentration of INCB018424.
Pharmacokinetics Parameter: AUC 0-12 of INCB018424 | Up to 24 weeks
  Defined as the area under the plasma or serum concentration-time curve from Hour 0 to 12 hours of INCB018424.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (22):
- United States (22):
  - Saguaro Dermatology, Phoenix, Arizona
  - First Oc Dermatology, Fountain Valley, California
  - Amicis Research Center Valencia, Northridge, California
  - Children'S Hospital of Orange County, Orange, California
  - Clinical Trials Research Institute, Thousand Oaks, California
  - Clarity Dermatology, Castle Rock, Colorado
  - International Clinical Research Tennessee Llc, Sanford, Florida
  - Lenus Research Medical Group, Llc, Sweetwater, Florida
  - Trueblue Clinical Research, Tampa, Florida
  - Lane Dermatology and Dermatologic Surgery, Columbus, Georgia
  - Options Research Group, Llc, West Lafayette, Indiana
  - Equity Medical, Llc, Bowling Green, Kentucky
  - Delricht Research, Baton Rouge, Louisiana
  - Revival Research Institute, Llc Troy, Troy, Michigan
  - Red River Research Partners, Bolivar, Missouri
  - Dr Bobby Buka, Md Greenwich Village, New York, New York
  - Equity Medical, Llc, New York, New York
  - Red River Research Partners, Fargo, North Dakota
  - Centricity Research Columbus, Columbus, Ohio
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - Paddington Testing Co Inc, Philadelphia, Pennsylvania
  - Dermresearch, Inc., Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study to Evaluate the Maximal Use of Ruxolitinib Cream in Adult and Adolescent Participants With Hidradenitis Suppurativa — https://www.incyteclinicaltrials.com/trials/INCB018424-112